CLINICAL TRIAL: NCT05964296
Title: Study of Impact on Therapeutic Alliance in People With Addiction Using the MAURISSE Application.
Brief Title: The Impact of the Use of the MAURISSE Application in People Suffering From an Addiction.
Acronym: ALMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/21/0540
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Substance Related Disorder; Personality Disorders
Keywords: eHealth; mHealth; application; substance use disorders; personality disorders; care observance; therapeutic alliance
MeSH Terms: conditions — Substance-Related Disorders; Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application group (Experimental): Patients randomized to the digital application arm will benefit from treatment as usual and will have access to the MAURISSE application, allowing them to communicate with the healthcare team using a messaging system, to report and follow substance use, to access a To-do list, to access personal multimedia contents helping with the treatment, to report a feeling of boredom (these moments presenting a risk of relapse) and finally to access a list of propositions in order to fight this feeling
  Interventions: Other: The MAURISSE application use
- Standard-of-care group (Active Comparator): These patients will benefit from the usual care within the center (appointments with doctors; regular follow-up meetings with nurses, psychologists, social workers, therapeutic groups depending on the evaluation).
  Interventions: Other: Usual care

INTERVENTIONS:
Other: The MAURISSE application use — * Exchanges with the care team via the messaging system,
  * Postponement of consumption,
  * Monitoring of consumption,
  * Access to information on the To Do List,
  * Access to personal content to help with management (Socio-professional situation, type of life, personal history..).
  * Postponement of a feeling of boredom,
  * Access to proposals to fight against this feeling.
  Arms: Application group
Other: Usual care — The usual care within the center will consist of appointments with doctors; regular follow-up meetings with nurses, psychologists, social workers, therapeutic groups depending on the evaluation.
  Arms: Standard-of-care group

SUMMARY:
Substance Use Disorders (SUD) are associated with cognitive schemas that lead to care attrition and mistrust towards care. Considering this, establishing a strong, trustful relationship between the patient and the healthcare team is important to promote patient engagement within SUD management. However, it requires an important availability of the healthcare team, allowing for frequent interactions at all times, including at night and during days off. We postulated that a mobile application called MAURISSE, which aims to help the caregivers maintaining a link with the patient in order to facilitate trust in the relationship, could foster patient engagement as well as the therapeutic alliance.

This research aims to compare the effect of the application MAURISSE on the therapeutic alliance in a population of patients treated for a disorder related to substance use at the Toulouse University Hospital.

DETAILED DESCRIPTION:
Substance Use Disorders (SUD) are frequently associated with other mental disorders, especially Borderline Personality Disorder, thus defining co-occurring substance use and mental disorders with borderline and anti-social personality disorders that is often associated with cognitive schemas leading to care attrition and mistrust towards care. The goal of the care intervention within Substance Use Disorders management is therefore to help the patient reduce the use of dysfunctional coping strategies involving substance use. Indeed, the establishment of a trustful relation between the patient and the care team leads the patient into building a secure attachment towards care that could secondly be generalized in other situations. We designed an application called MAURISSE, which aims to help the caregivers maintaining a link with the patient in order to facilitate a more secure attachment, thus enabling trust in the relationship as well as fostering patient engagement in the care.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old,
* Starting specialized treatment for addiction (addiction to substance and behavioral addiction too as money games addiction).
* Suffering from any type of addiction, with an active addiction requiring weekly monitoring of substance use.
* possessing a smartphone or having access to a smartphone and having access to an internet connection.
* Able to read and understand French.
* Affiliated or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patient with cognitive or psychiatric disorders that may affect their ability to consent.
* Participation in another protocol involving a modification of the treatment for addiction.
* Known or suspected pregnancy.
* Person under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The therapeutic alliance score assessed by the Working Alliance Inventory Short Revised scale (WAI-SR). | 2 months
  The Working Alliance Inventory-Short Revised is a scale that consists of two questionnaires. A 12-question questionnaire for patients and a 10-question questionnaire for caregivers. The questions are scored using a Likert scale ranging from 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Juliette SALLES, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France